CLINICAL TRIAL: NCT01039129
Title: Hybrid Transvaginal-Transabdominal Endoscopic Surgery
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit participants
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLR IRB#09-136
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2015-08-21 (Estimated); Status verified 2015-08

CONDITIONS: Gallstones; Appendicitis; Pelvic Pain
Keywords: Gallstones; Appendicitis; Pelvic pain; Peritoneal mass
MeSH Terms: conditions — Gallstones; Appendicitis; Pelvic Pain | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Endoscopic Cholecystectomy (Experimental): 20 patients in this arm will undergo cholecystectomy, or removal of the gallbladder, through this experimental approach. This arm will compose of patients with symptomatic gallstones (cholelithiasis).
  Interventions: Procedure: Endoscopic Cholecystectomy
- Endoscopic Appendectomy (Experimental): Participants will with chronic appendicitis will undergo appendectomy through this experimental approach.
  Interventions: Procedure: Endoscopic Appendectomy
- Endoscopic Peritoneoscopy (Experimental): 20 patients in this arm will undergo diagnostic peritoneoscopy with or without biopsy for any indication.
  Interventions: Procedure: Endoscopic Peritoneoscopy

INTERVENTIONS:
Procedure: Endoscopic Cholecystectomy — An incision will be made in the vagina and a flexible surgical camera (endoscope) and instruments will be introduced. The surgical procedure for each given arm will be performed with the aid of an additional surgical instrument inserted through a small incision in the umbilicus.
  Arms: Endoscopic Cholecystectomy
Procedure: Endoscopic Appendectomy — An incision will be made in the vagina and a flexible surgical camera (endoscope) and instruments will be introduced. The surgical procedure for each given arm will be performed with the aid of an additional surgical instrument inserted through a small incision in the umbilicus
  Arms: Endoscopic Appendectomy
Procedure: Endoscopic Peritoneoscopy — A diagnostic peritoneoscopy with or without biopsy for any indication
  Arms: Endoscopic Peritoneoscopy

SUMMARY:
The is a pilot study to evaluate the safety and efficacy of hybrid transvaginal-transabdominal procedures. Diagnostic peritoneoscopy (visualizing the inside of the abdomen), appendectomy (removal of the appendix), and cholecystectomy (removal of the gallbladder) will be performed through a vaginal incision with an additional small incision in the umbilicus.

ELIGIBILITY:
Inclusion Criteria:

* Chronic or early appendicitis
* Symptomatic gallstones
* Suspicious abdominal mass/nodule
* Female
* Age 18-60 years
* ASA Class I or II

Exclusion Criteria:

* Pregnant women
* History of previous abdominal, pelvic, or vaginal surgery
* History of previous abdominal or pelvic radiation therapy
* History of fibroid uterus
* History of endometriosis
* History of large ovarian cyst
* History of unexplained vaginal bleeding or dyspareunia

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2009-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Technical success | intra-operative
Complication | 1 month

SECONDARY OUTCOMES:
Operative time | intra-operative
Sexual function | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Julio Teixeira, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center, Department of Surgery
Locations (1):
- St. Luke's-Roosevelt Hospital Center, New York, New York, United States